CLINICAL TRIAL: NCT00963430
Title: A Phase II Study in Pregnant Women to Assess the Safety and Immunogenicity of an Unadjuvanted Sanofi Pasteur H1N1 Inactivated Influenza Vaccine Administered at Two Dose Levels
Brief Title: H1N1 Vaccine in Pregnant Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 09-0056; N01AI80004C
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Results first posted 2011-05-16 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2010-04

CONDITIONS: Influenza
Keywords: H1N1, influenza A viruses, pregnant women
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Group 2: 30 mcg H1N1 vaccine (Experimental): 60 subjects to receive 30 mcg of inactivated H1N1 vaccine on Day 0 and Day 21.
  Interventions: Biological: Inactivated H1N1 Vaccine
- Group 1: 15 mcg H1N1 vaccine (Experimental): 60 subjects to receive 15 mcg of inactivated H1N1 vaccine on Day 0 and Day 21.
  Interventions: Biological: Inactivated H1N1 Vaccine

INTERVENTIONS:
Biological: Inactivated H1N1 Vaccine — Two doses of inactivated influenza H1N1 vaccine delivered intramuscularly (IM) as 15 or 30 mcg dose. The 15 mcg dose will be administered as a single 0.5 mL IM injection in the deltoid muscle of the preferred arm. The 30 mcg dose will be administered as a single 1.0 mL injection in the deltoid muscle.

SUMMARY:
The purpose of this study is to evaluate an investigational 2009 H1N1 influenza vaccine to determine vaccine safety in pregnant women and the body's immune response (body's defense against disease) to different strengths of the H1N1 influenza vaccine. In this study, 2 strengths of the H1N1 influenza vaccine will be tested (given 3 weeks apart). Participants will include approximately 120 healthy pregnant women, ages 18-39 years, in their second or third trimester of pregnancy (14-34 weeks gestation). Study procedures will include 2 doses of vaccine, blood samples, cord blood samples at delivery, and recording temperature and vaccine side effects in a memory aid for 8 days following each vaccination. Participants will be involved in study related procedures for about 7 months.

DETAILED DESCRIPTION:
Recently, a novel swine-origin influenza A/H1N1 virus was identified as a significant cause of febrile respiratory illnesses in Mexico and the United States. It rapidly spread to many countries around the world, prompting the World Health Organization to declare a pandemic on June 11, 2009. Data from several cohorts in different age groups that received licensed trivalent seasonal influenza vaccines suggest that these vaccines are unlikely to provide protection against the new virus. In addition, adults are more likely to have measurable levels of serum hemagglutination inhibition assay (HAI) or neutralizing antibody than are children. These data indicate the need to develop vaccines against the new H1N1 strain and suggest that different vaccine strategies (e.g., number of doses, need for adjuvant) may be appropriate for persons in different age groups. Pregnant women are at an increased risk for the complications of influenza. A higher dose or multiple doses of an unadjuvanted, inactivated influenza H1N1 vaccine may be necessary to confer protection to this at risk population. This protocol will explore the antibody response following vaccination of pregnant women at 2 different dose levels (15 mcg and 30 mcg). The 2 doses of inactivated influenza H1N1 vaccine will be administered 21 days apart. This study will assess the immune response following a single dose of H1N1 vaccine, to assess whether individuals have any pre-existing "prime" immunity, such that the initial H1N1 vaccination serves as a boost, thus conferring a more rapid time to protection with the need for fewer doses. Antibody responses will be assessed 21 days after each dose. The primary objectives are: safety, to assess the safety of unadjuvanted, inactivated H1N1influenza vaccine in pregnant women when administered at the 15 mcg or 30 mcg dose; and immunogenicity, to assess the antibody response following a single dose of unadjuvanted, inactivated H1N1 influenza vaccine in pregnant women when administered at the 15 mcg or 30 mcg dose. The secondary objectives are to: assess the antibody response following 2 doses of unadjuvanted, inactivated H1N1 influenza vaccine in pregnant women when administered at the 15 mcg or 30 mcg dose; and assess the efficiency of placental transport of maternal influenza antigen specific antibodies to the neonate. This is a randomized, double-blinded, phase II study in 120 pregnant women, ages 18-39 years. Subjects will be randomized into 2 groups (60 pregnant women per dose group) to receive intramuscular inactivated influenza H1N1 vaccine at 15 mcg (Group 1) or 30 mcg (Group 2) on Days 0 and 21. Following immunization, safety will be measured by assessment of adverse events through 21 days following the last vaccination (Day 42), serious adverse events and new-onset chronic medical conditions through 7 months post first vaccination (Day 201). Reactogenicity to the vaccine will be assessed for 8 days following each vaccination (Day 0-7). Immunogenicity testing will include HAI and neutralizing antibody testing on serum obtained on Days 0, 21 and 42. This includes samples collected prior to each vaccination and samples collected 21 days following each vaccination. HAI antibody testing will be also be performed on serum from maternal and cord blood collected at delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant female between the ages of 18 and 39 years, inclusive.
* Is from 14-34 weeks of gestation, inclusive.
* Had at least one prenatal visit during which pregnancy was confirmed.
* Is in good health, as determined by vital signs (heart rate 100 beats per minute; blood pressure: systolic 140 mm Hg; diastolic less than or equal to 90 mm Hg; oral temperature less than 100 degrees Fahrenheit), medical history to ensure any existing medical diagnoses or conditions are stable and not considered clinically significant, and targeted physical examination based on medical history. A stable medical condition is defined as health outcomes of the specific disease are considered to be within acceptable limits in the last 3 months.
* Able to understand and comply with planned study procedures.
* Provides written informed consent prior to initiation of any study procedures.
* Agrees to sign medical release for herself and her infant(s) to allow study staff to gather pregnancy outcome data, if needed per clinical site policy.

Exclusion Criteria:

* Has a known allergy to eggs or other components in the vaccines (these may include, but are not limited to: gelatin, formaldehyde, octoxinol and chicken protein).
* Has a history of severe reactions following previous immunization with influenza virus vaccines.
* Has participated in a novel influenza H1N1 2009 vaccine study in the past 2 years or has history of novel influenza H1N1 2009 infection prior to enrollment.
* Has received any other live licensed vaccines within 4 weeks or inactivated licensed vaccines within 2 weeks prior to vaccination in this study prior to vaccination or plan receipt of such vaccines within 21 days following the last vaccination (except for seasonal inactivated influenza vaccine which may be received 2 weeks post either vaccination). Measles, mumps, and rubella vaccine and tetanus, diphtheria, and acellular pertussis vaccine are permitted post-partum.
* Has received an experimental/investigational agent (vaccine, drug, biologic, device, blood product, or medication) within one month prior to vaccination in this study, or expects to receive another experimental/investigational agent during the study period (prior to the Day 201 follow-up call - 180 days after the second vaccination).
* Has an acute illness and/or an oral temperature greater than or equal to 100.0 degrees Fahrenheit, within 72 hours of vaccination (This may result in a temporary delay of vaccination).
* Has immunosuppression as a result of an underlying illness or treatment, or use of anti-cancer chemotherapy or radiation therapy within the preceding 36 months.
* Has an active neoplastic disease (excluding non-melanoma skin cancer), a history of any hematologic malignancy, current bleeding disorder, or taking anticoagulants.
* Long term use of glucocorticoids, including oral or parenteral, or high-dose inhaled steroids (>800 micrograms/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (nasal and topical steroids are allowed) or has received betamethasone or dexamethasone to accelerate fetal lung maturity.
* Has a history of receiving immunoglobulin or other blood product (with exception of Rhogam) within the 3 months prior to enrollment in this study.
* Has a diagnosis of a current and uncontrolled major psychiatric disorder.
* Has been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others, within the past 10 years.
* The subject is receiving any of the following psychiatric drugs: aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, trifluopromazine, chlorprothixene, chlorpromazine, perphenazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate. Subjects who are receiving an antidepressant drug (not listed above) and are stable for at least 3 months prior to enrollment without decompensating are allowed enrollment into the study.
* Known active human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infection.
* History of alcohol or drug abuse in the last 5 years.
* Has a seizure disorder or is on an anti-seizure medication.
* Has a history of Guillain-Barré Syndrome.
* Plan to travel outside of North America in the time between the first vaccination and 42 days following the first vaccination.
* Has an acute or chronic medical condition that, in the opinion of the investigator would render vaccination unsafe, or would interfere with the evaluation of responses (this includes, but is not limited to, known cardiac disease, chronic liver disease, significant renal disease, unstable or progressive neurological disorder, transplant recipients or uncontrolled diabetes, juvenile diabetes (Type I) or advanced diabetes with renal disease or eye disease, diabetes controlled by diet or insulin is acceptable.)
* Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2009-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Saint Louis University - Center for Vaccine Development, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine - Department of Molecular Virology and Microbiology, Houston, Texas
  - Group Health Cooperative, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy pregnant women recruited from existing volunteer populations and from the communities at large around the clinical sites. Participants were enrolled between 09Sep2009 and 16Oct2009.
Groups:
- 15 Mcg H1N1 Vaccine: Participants received 15 mcg of Inactivated H1N1 Vaccine by intramuscular injection on Day 0 and Day 21.
- 30 Mcg H1N1 Vaccine: Participants received 30 mcg of Inactivated H1N1 Vaccine by intramuscular injection on Day 0 and Day 21.
Period: Overall Study
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Started | 60 | 60
Completed | 59 | 57
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 60 | 120
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 31.7 (4.3) | 31.2 (4.3) | 31.4 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 60 | 120
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Solicited Subjective Local Reactions After First Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of local reactions of pain, tenderness and swelling for 8 days after vaccination (Day 0-7) based on their interference with daily activities. Participants are counted if they were reported as experiencing the symptom at any severity on any of the 8 days.
Time Frame: Within 8 days (Day 0-7) post first vaccination
Population: All participants receiving the first vaccination are included in the safety cohort. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 60 | 60
Participants
  Pain | 15 | 21
  Tenderness | 26 | 37
  Swelling | 1 | 1

2. Primary Outcome: Number of Participants Reporting Solicited Subjective Local Reactions After Second Vaccination
Description: as for outcome 1
Time Frame: Within 8 days (Day 0-7) post second vaccination
Population: All participants receiving the second vaccination are included in the safety cohort. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 49 | 54
Participants
  Pain | 10 | 20
  Tenderness | 26 | 37
  Swelling | 1 | 0

3. Primary Outcome: Number of Participants Reporting Solicited Quantitative Local Reactions After First Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of local reactions of redness and swelling for 8 days after vaccination (Day 0-7). If the reaction was present, the maximum diameter was measured in millimeters (mm). Participants are counted if they reported experiencing the reaction with any measurement greater than 0 mm on any of the 8 days.
Time Frame: Within 8 days (Day 0-7) post first vaccination
Population: All participants receiving the first vaccination are included in the safety cohort. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 60 | 60
Participants
  Redness | 5 | 8
  Swelling | 4 | 1

4. Primary Outcome: Number of Participants Reporting Solicited Quantitative Local Reactions After Second Vaccination
Description: as for outcome 3
Time Frame: Within 8 days (Day 0-7) post second vaccination
Population: All participants receiving the second vaccination are included in the safety cohort. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 49 | 54
Participants
  Redness | 2 | 3
  Swelling | 1 | 0

5. Primary Outcome: Number of Participants Reporting Solicited Subjective Systemic Reactions After First Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of systemic symptoms of feverishness, malaise, myalgia, headache, and nausea for 8 days after vaccination (Day 0-7) based on their interference with daily activities. Participants are counted if they reported experiencing the symptom at any severity on any of the 8 days.
Time Frame: Within 8 days (Day 0-7) post first vaccination
Population: All participants receiving the first vaccination are included in the safety cohort. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 60 | 60
Participants
  Feverishness | 5 | 4
  Malaise | 19 | 24
  Myalgia | 12 | 8
  Headache | 17 | 18
  Nausea | 10 | 12

6. Secondary Outcome: Number of Participants With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer Greater Than or Equal to 40 Against the Novel Influenza H1N1 2009 Virus in the Maternal Blood at the Time of Delivery
Description: Blood was collected from participants at the time of delivery for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: At time of delivery
Population: Participants were included in the analyses if they had blood collected at delivery, with 22 participants excluded due to receipt of non-study vaccines and 3 due to specimen processing errors at the time of sample collection. Participants were analyzed as treated.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 41 | 47
Participants | 35 | 29

7. Secondary Outcome: Number of Participants With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer Greater Than or Equal to 40 Against the Novel Influenza H1N1 2009 Virus in Cord Blood
Description: Cord blood was collected at the time of delivery for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: At time of delivery
Population: Participants were included in the analyses if a cord blood sample was collected at delivery, with 22 participants excluded due to receipt of non-study vaccines and 5 due to specimen processing errors at the time of sample collection.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 39 | 46
Participants | 34 | 41

8. Secondary Outcome: Number of Participants With 4-fold or Greater Serum Hemagglutination Inhibition (HAI) Antibody Titer Increases Against Influenza H1N1 2009 Virus Following 2 Doses of H1N1 Vaccine
Description: Blood was collected from all participants prior to the initial vaccination as well as 21 days after the second vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 21 post vaccination 2 titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 21 post vaccination 2 titer was an increase by 4-fold or more.
Time Frame: Day 0 prior to first vaccination and Day 21 after the second vaccination
Population: Participants were included in the analyses if they received both vaccinations within 4 days of the window and had blood collected at both timepoints, with 13 participants excluded due to receipt of non-study vaccines. Participants were analyzed as treated.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 38 | 51
Participants | 36 | 47

9. Primary Outcome: Number of Participants Reporting Solicited Subjective Systemic Reactions After Second Vaccination
Description: as for outcome 5
Time Frame: Within 8 days (Day 0-7) post second vaccination
Population: All participants receiving the second vaccination are included in the safety cohort. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 49 | 54
Participants
  Feverishness | 2 | 4
  Malaise | 8 | 14
  Myalgia | 3 | 6
  Headache | 11 | 11
  Nausea | 2 | 4

10. Primary Outcome: Number of Participants Reporting Fever After First Vaccination
Description: Participants were provided with a thermometer and a memory aid on which to record daily oral temperatures for 8 days after vaccination (Day 0-7). The protocol defined fever as oral temperature of 37.8 degrees Celsius or higher. Participants are counted as experiencing fever if they reported oral temperatures of 37.8 degrees Celsius or higher on any of the 8 days.
Time Frame: Within 8 days (Day 0-7) post first vaccination
Population: All participants receiving the first vaccination are included in the safety cohort. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 60 | 60
Participants | 0 | 1

11. Primary Outcome: Number of Participants Reporting Fever After Second Vaccination
Description: as for outcome 10
Time Frame: Within 8 days (Day 0-7) post second vaccination
Population: All participants receiving the second vaccination are included in the safety cohort. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 49 | 54
Participants | 1 | 0

12. Primary Outcome: Number of Participants With 4-fold or Greater Serum Hemagglutination Inhibition (HAI) Antibody Titer Increases Against Influenza H1N1 2009 Virus Following a Single Dose of H1N1 Vaccine
Description: Blood was collected from all participants prior to the initial vaccination as well as 21 days after the first vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 21 post vaccination titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 21 post vaccination titer was an increase by 4-fold or more.
Time Frame: Day 0 prior to and Day 21 after the first vaccination
Population: Participants were included in the analyses if they received the first vaccination and had blood collected at both timepoints, with 5 participants excluded due to receipt of non-study vaccines. Participants were analyzed as treated.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 55 | 58
Participants | 49 | 56

13. Primary Outcome: Number of Participants With a Serum Hemagglutination Inhibition (HAI) Antibody Titer of 1:40 or Greater Against Influenza H1N1 2009 Virus Following a Single Dose of H1N1 Vaccine
Description: Blood was collected from all participants at Day 21 post first vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 21 after the first vaccination
Population: Participants were included in the analyses if they received the first vaccination and had blood collected at the timepoint, with 5 participants excluded due to receipt of non-study vaccines. Participants were analyzed as treated.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 55 | 58
Participants | 51 | 56

14. Primary Outcome: Number of Participants Reporting Maternal Complications of Pregnancy, Labor and Delivery
Description: Participants were contacted after delivery, and medical records reviewed, to collect complications experienced during pregnancy, labor and delivery. The data collection process followed a prospectively-defined list of complications reported for this outcome measure, some of which may have also been reported as serious adverse events if otherwise meeting those requirements.
Time Frame: At time of delivery
Population: All participants from whom outcome data were collected are included in the ITT safety population for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 60 | 60
Participants
  Stillborn | 1 | 0
  Miscarriage | 1 | 0
  Gestational diabetes | 1 | 4
  Polyhydramnios | 1 | 0
  Oligohydramnios | 2 | 2
  Pregnancy induced hypertension | 0 | 3
  Pre-eclampsia | 1 | 2
  Eclampsia | 0 | 0
  Fetal Distress | 1 | 3
  Abruptio Placenta | 1 | 0
  Chorioamnionitis | 3 | 2
  Fever | 2 | 2
  Anaphylaxis | 0 | 0
  Antibiotics prior to delivery | 26 | 20
  Fetal abnormalities detected during pregnancy | 3 | 5
  Assisted vaginal delivery | 4 | 3
  Non-elective Cesarean section | 4 | 4
  Abnormal amniotic fluid | 11 | 12
  Postpartum fever | 1 | 0
  Postpartum endometritis | 0 | 0
  Postpartum bleeding | 5 | 5
  Postpartum bacteremia | 0 | 0

15. Primary Outcome: Number of Participants Reporting Neonatal Complications
Description: Participants were contacted after delivery, and medical records reviewed, to collect neonatal complications. The data collection process followed a prospectively-defined list of complications reported for this outcome measure, some of which may have also been reported as serious adverse events if otherwise meeting those requirements.
Time Frame: At time of delivery
Population: All live births are included in this outcome measure, which excludes 2 participants whose pregnancies ended in miscarriage or stillbirth. Three participants gave birth to twins and one to triplets, each counted separately.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 61 | 62
Participants
  Pre-term (less than 37 weeks) | 10 | 7
  Large for gestational age | 12 | 3
  Small for gestational age | 3 | 1
  Abnormal infant exam | 15 | 13
  Congenital abnormalities | 1 | 3
  Hematological complications | 3 | 1
  Infection | 0 | 0
  Sepsis | 0 | 0
  Meningitis | 0 | 0
  Metabolic complications | 4 | 0
  Respiratory complications | 6 | 3
  Respiratory support used | 5 | 3
  Fever 100.4 degrees Fahrenheit or greater | 0 | 0
  Admission to special nursery/infant intensive care | 6 | 6

16. Secondary Outcome: Number of Participants With a Serum Hemagglutination Inhibition (HAI) Antibody Titer of 1:40 or Greater Against Influenza H1N1 2009 Virus Following 2 Doses of H1N1 Vaccine
Description: Blood was collected from all participants at Day 21 post second vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 21 after the second vaccination
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 38 | 51
Participants | 36 | 47

17. Primary Outcome: Number of Participants Reporting Vaccine-associated Serious Adverse Events (SAEs)
Description: Serious adverse events included any untoward medical occurrence that resulted in death of the mother, fetus or infant; was life threatening to mother, fetus or infant; was a persistent/significant disability/incapacity; required in-patient hospitalization or prolongation thereof; was a congenital anomaly/birth defect in fetus or infant; or may have jeopardized the mother, fetus or infant, or required intervention to prevent one of the outcomes, or was described as Guillain-Barré Syndrome. Association was determined by a clinician licensed to diagnose and listed on the site's FDA Form 1572.
Time Frame: Day 0 through Day 180 after last vaccination
Population: All participants receiving the first vaccination are included in the ITT safety cohort.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 60 | 60
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited events were collected for 8 days after each vaccination, unsolicited events through 21 days after last vaccination, and serious adverse events and new onset chronic medical conditions through 180 days after last vaccination.
Description: For events solicited on a Memory Aid in the 8 days after vaccination, a participant was considered to have one event if it was reported as experienced at any time in the 8 day period.
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Serious Adverse Events (participants affected / at risk) | 9/60 | 6/60
Other Adverse Events (participants affected / at risk) | 53/60 | 54/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 Mcg H1N1 Vaccine (N=60) | 30 Mcg H1N1 Vaccine (N=60)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 2 (2)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Myomectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Caesarean section (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
HELLP syndrome (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Pregnancy induced hypertension (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 Mcg H1N1 Vaccine (N=60) | 30 Mcg H1N1 Vaccine (N=60)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 10 (11)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3)
Feeling hot (General disorders) | 7 (7) | 8 (8)
Malaise (General disorders) | 23 (27) | 28 (38)
Myalgia (Musculoskeletal and connective tissue disorders) | 15 (15) | 11 (14)
Headache (Nervous system disorders) | 23 (28) | 24 (29)
Nausea (Gastrointestinal disorders) | 10 (12) | 14 (16)
Injection site pain (General disorders) | 21 (25) | 31 (41)
Tenderness (General disorders) | 37 (52) | 44 (74) — Tenderness was solicited as a reaction at the vaccination site.
Injection site erythema (General disorders) | 6 (7) | 9 (11)
Injection site swelling (General disorders) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less